CLINICAL TRIAL: NCT02261883
Title: Intravenous Remodulin (Treprostinil) as Add-on Therapy for the Treatment of Persistent Pulmonary Hypertension of the Newborn: A Randomized, Placebo-Controlled, Safety and Efficacy Study
Brief Title: Remodulin as Add-on Therapy for the Treatment of Persistent Pulmonary Hypertension of the Newborn
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIV-PN-201
Record Dates: First submitted 2013-10-30; First posted 2014-10-10 (Estimated); Results first posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Persistent Pulmonary Hypertension of the Newborn
Keywords: PPHN
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome | interventions — treprostinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IV Remodulin (Active Comparator): The starting dose was 1 ng/kg/min (not to exceed to 2 ng/kg/min) and was titrated by up to 2 ng/kg/min every 2 hours, as tolerated and clinically indicated by the Investigator. Doses were titrated and maximized throughout the study until the desired clinical effect was observed or to each individual subject's maximally tolerated dose. There was no maximum dose.
  Interventions: Drug: IV Remodulin
- Placebo (Placebo Comparator): The starting dose was 1 ng/kg/min (not to exceed to 2 ng/kg/min) and was titrated by up to 2 ng/kg/min every 2 hours, as tolerated and clinically indicated by the Investigator. Doses were titrated and maximized throughout the study until the desired clinical effect was observed or to each individual subject's maximally tolerated dose. There was no maximum dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IV Remodulin — Treprostinil is a chemically stable tricyclic analogue of prostacyclin.
  Other Names: Treprostinil
  Arms: IV Remodulin
Drug: Placebo — Sodium citrate, sodium chloride, sodium hydroxide pellets, metacresol, and citric acid (anhydrous).
  Arms: Placebo

SUMMARY:
This study assessed the safety and treatment effect of intravenous (IV) Remodulin as an add-on therapy in neonates with persistent pulmonary hypertension of the newborn (PPHN).

DETAILED DESCRIPTION:
This study was designed to investigate if the addition of Remodulin reduced the rate of clinical worsening (defined as the need for additional treatment targeting PPHN, need for extracorporeal mechanical oxygenation [ECMO], or death) in neonatal subjects with PPHN who did not show an adequate response to inhaled nitric oxide (iNO). This study was part of a pediatric investigation plan agreed upon by the EMA (EMEA 000207-PIP01-08-M08).

ELIGIBILITY:
Inclusion Criteria:

* Parent(s) or legal guardian provided consent for the subject to participate
* Weight at least 2 kg at Screening
* Gestational age of ≥34 weeks and ≤14 days old at Screening
* Diagnosis of PPHN, which was either idiopathic in nature or associated with the following: meconium aspiration syndrome, pneumonia, respiratory distress syndrome, sepsis, birth hypoxia, perinatal encephalopathy, or unilateral congenital diaphragmatic hernia
* Currently requiring ventilator support
* Two consecutive oxygenation index (OI) of 15 or greater separated by at least 30 minutes, after receiving iNO for at least 3 hours
* Echocardiographic (ECHO) evidence of pulmonary hypertension with elevated right ventricle pressure
* Dedicated venous access for the administration of study drug (central line or peripherally inserted central venous catheter)

Exclusion Criteria:

* Previous or concurrent use of a phosphodiesterase-5 inhibitor, endothelin receptor antagonist, or prostanoid
* Significant congenital heart disease as detected by ECHO, minor valvular abnormalities, or expected transitional findings such as a patent foramen ovale, or patent ductus arteriosus.
* Clinically significant, untreated active pneumothorax at Screening
* Evidence of clinically significant bleeding at Screening
* Necrotizing enterocolitis (≥Bells stage II at Screening)
* Uncontrolled hypotension (mean systemic pressures ≤35 mmHg at Screening)
* Uncontrolled coagulopathy and / or untreated thrombocytopenia (<50,000 platelets/µL at Screening)
* History of severe (Grade 3 or 4) intracranial hemorrhage at Screening
* Currently receiving extracorporeal mechanical oxygenation (ECMO) or had immediate plans to initiate ECMO
* Expected duration on mechanical ventilation of <48 hours
* Life expectancy was less than 2 months or had a lethal chromosomal anomaly
* Contraindication to ECMO
* Bilateral congenital diaphragmatic hernia
* Active seizures at Screening
* Currently participating in another clinical drug study

Ages: 1 Hour to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2015-07-29 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2023-05-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Stanford Children's Hospital, Palo Alto, California
  - All Children's Hospital, St. Petersburg, Florida
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Mississippi Medical Center - Baston Children's Hospital, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Columbia University Medical Center, New York, New York
  - Nationwide Childrens Hospital, Columbus, Ohio
  - Cook Children's Medical Center, Fort Worth, Texas
  - University of Virginia Health Systems (UVA), Charlottesville, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Wauwatosa, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IV Remodulin | Placebo
Started | 21 | 21
Completed | 15 | 18
Not Completed | 6 | 3
Not completed — Death | 3 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Required ECMO Prior to Study Drug Administration | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population
Groups:
- Placebo: The starting dose was 1 ng/kg/min (not to exceed to 2 ng/kg/min) and was titrated by up to 2 ng/kg/min every 2 hours, as tolerated and clinically indicated by the Investigator. Doses were titrated and maximized throughout the study until the desired clinical effect was observed or to each individual subject's maximally tolerated dose. There was no maximum dose.
  Placebo: Sodium citrate USP/EP/JP, sodium chloride USP/EP/JP, sodium hydroxide pellets, metacresol, and citric acid (anhydrous).
- Total: Total of all reporting groups
Arm/Group | IV Remodulin | Placebo | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Median (Full Range); unit: days] | 2.0 [1 to 6] | 3.0 [1 to 6] | 3.0 [1 to 6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 10 | 11 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 17 | 19 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 10 | 15
  White | 12 | 11 | 23
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Gestational Age [Median (Full Range); unit: weeks] | 39.00 [34.0 to 41.0] | 39.00 [34.0 to 41.2] | 39.00 [34.0 to 41.2]
Birth Weight [Median (Full Range); unit: kg] | 3.08 [2.2 to 4.8] | 3.06 [2.2 to 4.5] | 3.06 [2.2 to 4.8]
Oxygenation Index [Median (Full Range); unit: units on a scale] — OI is an assessment of how much oxygen from the lungs enters the blood when a subject inhales, calculated as: mean airway pressure (MAP) multiplied by fraction of inspired oxygen (FiO2) divided by partial pressure of oxygen in the arterial blood (PaO2), then multiplying by 100. An OI of 15 or less indicates mild hypoxia, 16 to 25 indicates moderate hypoxia, 26 to 40 indicates severe hypoxia, and more than 40 indicates very severe hypoxia.
  units on a scale | 25.5 [4 to 46] | 22.0 [6 to 46] | 23.0 [4 to 46]
Fraction of Inspired Oxygen (FiO2) [Median (Full Range); unit: percentage of oxygen] — FiO2 is the concentration of oxygen in the air that a person inhales. FIO2 is expressed as a fraction or percentage, indicating the proportion of inspired air that consists of oxygen. If a patient is on 100% oxygen, the FIO2 is 1.0, indicating that the inspired air consists of only oxygen. On the other hand, room air, which typically contains about 21% oxygen, corresponds to an FIO2 of 0.21.
  percentage of oxygen | 100.0 [75 to 100] | 100.0 [35 to 100] | 100.0 [35 to 100]
Partial Pressure of Oxygen (PaO2) [Median (Full Range); unit: mmHg] — PaO2 is a measure of the pressure exerted by oxygen molecules in the arterial blood. PaO2 is an important parameter used in blood gas analysis to assess the oxygenation status of a patient. A blood sample is taken from an artery to measure PaO2. PaO2 is typically reported in millimeters of mercury (mmHg) and reflects the partial pressure of oxygen dissolved in the arterial blood. Normal PaO2 levels can vary slightly depending on factors such as age, altitude, and individual health conditions. However, in general, normal arterial oxygen levels at sea level are around 80 to 100 mmHg.
  mmHg | 51.0 [33 to 153] | 57.0 [32 to 286] | 56.0 [32 to 286]
PaO2/FiO2 (P/F Ratio) [Median (Full Range); unit: ratio] — PaO2/FiO2 ratio, also referred to as P/F Ratio, is a calculation used to assess the severity of hypoxemia, which is a condition characterized by low levels of oxygen in the blood. A low P/F ratio suggests that the patient's oxygen levels are compromised relative to the amount of oxygen being provided.
  ratio | 0.57 [0.4 to 1.6] | 0.69 [0.4 to 2.9] | 0.60 [0.4 to 2.9]
Inhaled Nitric Oxide (iNO) [Median (Full Range); unit: ppm] — iNO is a medication administered through inhalation to help dilate blood vessels in the lungs, improve oxygenation, and reduce pulmonary hypertension. The amount of medication delivered is measured in parts per million (ppm) of the gas that the patient inhales.
  ppm | 20.00 [20.0 to 20.0] | 20.00 [20.0 to 20.0] | 20.00 [20.0 to 20.0]
N-terminal pro-B-type natriuretic peptide (NT-proBNP) [Median (Full Range); unit: pg/mL] — NT-proBNP is a biomarker used to assess heart function and identify certain cardiac conditions. It is a hormone released by the heart, specifically by the ventricles, in response to increased pressure or volume. Elevated levels of NT-proBNP in the blood generally indicate increased strain or stress on the heart.
  pg/mL | 11194.0 [792 to 31366] | 16646.0 [1011 to 70000] | 13628.0 [792 to 70000]
Time Since Diagnosis [Median (Full Range); unit: days] — The number of days since the subject was diagnosed with persistent pulmonary hypertension of the newborn (PPHN).
  days | 2.0 [1 to 6] | 2.0 [1 to 6] | 2.0 [1 to 6]
PPHN Diagnosis [Count of Participants; unit: Participants]
  Idiopathic PPHN | 0 | 1 | 1
  Associated with Meconium Aspiration Syndrome | 9 | 10 | 19
  Associated with Respiratory Distress Syndrome | 5 | 3 | 8
  Associated with Sepsis | 0 | 1 | 1
  Associated with Birth Hypoxia | 1 | 1 | 2
  Associated with Unilateral Congenital Diaphragmatic Hernia | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Experiencing Clinical Worsening
Description: Clinical worsening was a composite endpoint defined by the occurrence of 1 of the following: death, initiation of ECMO per institutional policies, or need for additional treatment (initiation of additional targeted pulmonary vasodilator therapy).
Time Frame: From Baseline to Day 14
Population: Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | IV Remodulin | Placebo
Number analyzed (Participants) | 20 | 21
Participants
  Yes | 8 | 12
  No | 12 | 9

2. Secondary Outcome: Change in Oxygenation Index (OI)
Description: OI is an assessment of how much oxygen from the lungs enters the blood when a subject inhales, calculated as: mean airway pressure (MAP) multiplied by fraction of inspired oxygen (FiO2) divided by partial pressure of oxygen in the arterial blood (PaO2), then multiplying by 100. An OI of 15 or less indicates mild hypoxia, 16 to 25 indicates moderate hypoxia, 26 to 40 indicates severe hypoxia, and more than 40 indicates very severe hypoxia.
Time Frame: From Baseline to Hours 12, 24, and 72; Days 7 and 14; and/or prior to study drug discontinuation/weaning
Population: Intent-to-Treat Population
Measure: Median (Full Range); unit: units on a scale
Arm/Group | IV Remodulin | Placebo
Number analyzed (Participants) | 20 | 21
units on a scale
  12 Hours | -2.0 [-41 to 37] | -3.5 [-29 to 34]
  24 Hours | -8.5 [-40 to 23] | -5.5 [-30 to 58]
  72 Hours | -7.0 [-40 to 65] | -10.0 [-41 to 83]
  Day 7 | -9.5 [-40 to 36] | -11.0 [-43 to 42]
  Day 14 | -12.0 [-40 to 36] | -14.0 [-35 to 42]

3. Secondary Outcome: Change in P/F Ratio
Description: PaO2/FiO2 ratio, also referred to as P/F Ratio, is a calculation used to assess the severity of hypoxemia, which is a condition characterized by low levels of oxygen in the blood. A low P/F ratio suggests that the patient's oxygen levels are compromised relative to the amount of oxygen being provided.
Time Frame: From Baseline to Hours 12, 24, and 72
Population: Intent-to-Treat Population
Measure: Median (Full Range); unit: ratio
Arm/Group | IV Remodulin | Placebo
Number analyzed (Participants) | 20 | 21
ratio
  12 Hours | 0.11 [-0.5 to 10.5] | 0.10 [-2.3 to 4.1]
  24 Hours | 0.35 [-0.4 to 9.3] | 0.27 [-2.3 to 7.1]
  72 Hours | 0.50 [-0.4 to 4.8] | 0.65 [-2.3 to 7.5]

4. Secondary Outcome: Change in Pre- and Post-ductal Oxygen Saturation (SpO2)
Description: SpO2 is an assessment of how much oxygen is in the blood, measured by a pulse oximeter. Pre-ductal SpO2 is measured in the right hand or foot and is a reflection of the amount of oxygen flowing to the brain. Post-ductal SpO2 is measured in the left hand or foot, after the blood has mixed with less oxygenated blood from the rest of the body.
Time Frame: From Baseline to Hours 6, 12, 24, and 72
Population: Intent-to-Treat Population
Measure: Median (Full Range); unit: percentage of oxygen
Arm/Group | IV Remodulin | Placebo
Number analyzed (Participants) | 20 | 21
percentage of oxygen
  6 Hours | 3.0 [-6 to 13] | 1.0 [-10 to 7]
  12 Hours | 3.0 [-7 to 17] | 0.5 [-7 to 12]
  24 Hours | 3.0 [-12 to 15] | 1.0 [-17 to 11]
  72 Hours | 0.0 [-4 to 16] | 1.5 [-21 to 8]

5. Secondary Outcome: Change in N-terminal Pro-Brain Natriuretic Peptide (NT-proBNP)
Description: NT-proBNP is a hormone produced by the heart. Increased NT-proBNP concentration is associated with changes in right heart morphology and function. The main purpose of NT-proBNP testing is to see if the blood levels of this protein are within the expected range for a healthy individual.
Time Frame: From Baseline to Days 1, 2, 3, 7, and 14 (or prior to hospital discharge)
Population: Intent-to-Treat Population
Measure: Median (Full Range); unit: pg/mL
Arm/Group | IV Remodulin | Placebo
Number analyzed (Participants) | 20 | 21
pg/mL
  Day 1 | -1577.00 [-21322.0 to 43388.0] | -1378.00 [-23206.0 to 17923.0]
  Day 2 | -1955.00 [-24637.0 to 34599.0] | -4090.00 [-37390.0 to 14163.0]
  Day 3 | -252.00 [-24623.0 to 30629.0] | -4090.00 [-49200.0 to 13550.0]
  Day 7 | 484.00 [-24623.0 to 19970.0] | -11312.00 [-65387.0 to 12299.0]
  Day 14 | -719.00 [-26283.0 to 56529.0] | -9003.00 [-65387.0 to 12299.0]

6. Secondary Outcome: Time to Clinical Worsening
Description: Clinical worsening was assessed continuously during the study. Clinical worsening was a composite endpoint defined by the occurrence of 1 of the following: death, initiation of ECMO per institutional policies, or need for additional treatment (initiation of additional targeted pulmonary vasodilator therapy).
Time Frame: From Baseline to Day 56
Population: Intent-to-Treat Population
Measure: Median (Full Range); unit: days
Arm/Group | IV Remodulin | Placebo
Number analyzed (Participants) | 8 | 12
days | 3.0 [1 to 8] | 3.0 [1 to 13]

7. Secondary Outcome: Time to Initiation of ECMO
Description: Start of ECMO was assessed continuously during the study. ECMO is a life-support therapy that oxygenates blood by passing it through an artificial lung. The start time of ECMO, if needed, was recorded for each subject.
Time Frame: From Baseline to Day 56
Population: Intent-to-Treat Population
Measure: Median (Full Range); unit: days
Arm/Group | IV Remodulin | Placebo
Number analyzed (Participants) | 6 | 7
days | 2.5 [1 to 8] | 3.0 [1 to 5]

8. Secondary Outcome: Time to Discontinuation of Inhaled Nitric Oxide (iNO)
Description: Discontinuation of iNO was assessed continuously during the study. iNO works by relaxing the blood vessels in the lungs, which makes it easier for oxygen to be delivered to the body. The stop time of iNO was recorded for each subject.
Time Frame: From Baseline to Day 56
Population: Intent-to-Treat Population
Measure: Median (Full Range); unit: days
Arm/Group | IV Remodulin | Placebo
Number analyzed (Participants) | 20 | 21
days | 7.5 [1 to 12] | 7.0 [1 to 11]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were captured from when the subject signed the informed consent form until the subject completed the study or was withdrawn from the study, up to 56 days.
Description: AEs were followed until either resolution (or return to normal or baseline values), until they were judged by the Investigator to no longer be clinically significant, or for at least 4 weeks after the last dose of study drug. All serious adverse events (SAEs) were followed until resolution, death, or the subject was lost to follow-up, even if they were ongoing more than 4 weeks after completion of the last dose of study drug.
Arm/Group | IV Remodulin | Placebo
All-Cause Mortality (participants affected / at risk) | 4/20 | 2/21
Serious Adverse Events (participants affected / at risk) | 8/20 | 3/21
Other Adverse Events (participants affected / at risk) | 19/20 | 17/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Remodulin (N=20) | Placebo (N=21)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Congenital diaphragmatic hernia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Remodulin (N=20) | Placebo (N=21)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Drug withdrawal syndrome neonatal (General disorders) | 3 (3) | 0 (0)
Drug withdrawal syndrome (General disorders) | 1 (1) | 2 (2)
Oedema (General disorders) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Hypotension (Vascular disorders) | 6 (7) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator agree not to publish or publicly present any results of the Study without the prior written consent of Sponsor, not to be unreasonably withheld or delayed. Institution and/or Principal Investigator further agree to provide Sponsor with drafts of any such publication or presentation for review and approval no less than 30 days prior to submission for publication or the date of public presentation.

DOCUMENTS (2):
  • Study Protocol (2016-04-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT02261883/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT02261883/SAP_001.pdf